CLINICAL TRIAL: NCT04153630
Title: Safety Study and Preliminary Efficacy of Infusion Haploidentical Mesenchymal Stem Cells Derived From Bone Marrow for Treating Recessive Dystrophic Epidermolysis Bullosa
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Universidad Carlos III Madrid (TERMeG) (Unknown); St John's Institute of Dermatology Kings College London (Unknown); Instituto de Salud Carlos III (Other Government); DEBRA (Unknown); CIBER Enfermedades raras (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MesenSistem-EB
Record Dates: First submitted 2019-08-06; First posted 2019-11-06 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-04

CONDITIONS: Epidermolysis Bullosa Dystrophica, Recessive
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Haploidentical MSCs derived from bone marrow (Experimental): Haploidentical MSCs derived from bone marrow administered by intravenous injection with a dose of 2-3x106 cells / Kg
  Interventions: Biological: mesenchymal stem cells derived from bone marrow (BM-MSCs)

INTERVENTIONS:
Biological: mesenchymal stem cells derived from bone marrow (BM-MSCs) — Procedure: Haploidentical MSCs derived from bone marrow administered by intravenous injection with a dose of 2-3x106 cells / Kg

SUMMARY:
Phase I / II pilot clinical trial, to evaluate the safety and preliminary efficacy of the systemic infusion of mesenchymal stem cells derived from bone marrow (BM-MSCs) from a haploidentical donor to improve the healing process and / or the mucocutaneous fragility phenotype associated with EBDR.

DETAILED DESCRIPTION:
The Main Objective is to evaluate the safety and therapeutic efficacy of haploidentical MSCs derived from bone marrow administered by intravenous injection for the treatment of patients with RDBS. The assessment of the symptomatic improvement of the treated patients will be made regarding the baseline situation and the response to treatment at the biochemical, histological and molecular level.

Secondary Objectives:

Describe the clinical and molecular phenotype of the mucocutaneous involvement of patients, including the characterization of the mutations responsible for the disease.

Study drug: Allogenic mesenchymal cells (haploidentical) derived from bone marrow and expanded.

Method of administration: Systemic / Intravenous Administration dose: 2-3x10e6 BM-MSC / Kg. Weekly dose for three consecutive weeks

Follow-up period: 12 months after the infusion. However, patients will be monitored outside the clinical trial over a 5-year period

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 12 months and ≤ 18 years of age at the time of inclusion in the study.
2. Patients with a clinical, molecular and genetic diagnosis of EBDR.
3. Patients with presence of the NC-1 domain of type VII collagen, in skin biopsies and/or Western-Blot, detected with a battery of specific antibodies.
4. Patients with a haploidentical donor.
5. Subjects with a severity score> 20 according to "The Birmingham Epidermolysis Bullosa Severity Score".
6. Minor subjects whose representative / legal guardian has voluntarily signed the informed consent before the first intervention of the study.
7. In the case of mature minors (12-17 years of age), in addition to the consent signed by the legal guardian, the consent of the minor will be obtained.
8. Women with reproductive capacity must have a negative pregnancy test at the time of inclusion and must agree to use highly effective contraceptive methods (diaphragms plus spermicide or male condom plus spermicide, oral contraceptive combined with a second method contraceptive implant, contraceptive injectable, permanent intrauterine device, sexual abstinence or partner with vasectomy) during their participation in the study until 30 days after the last visit.
9. Males should agree to use a double-barrier contraceptive method (condom plus spermicide or diaphragm plus spermicide) during their participation in the study and up to 30 days after the last dose of the study drug, or the male patient or his Female partners must be surgically sterilized or the female partner must be postmenopausal.
10. The patient must be able to attend all study visits and comply with all study procedures.

Exclusion Criteria:

1. Subjects who for medical reasons can not be moved to the University Hospital La Paz in Madrid.
2. Subjects who have received immunotherapy including oral corticosteroids (> 15 mg / day) for more than 1 week (excluding inhaled and ophthalmic preparations) or chemotherapy 8 days prior to inclusion in the study. The inclusion of the patient is understood from the signing of the informed consent.
3. Subjects with a known allergy to any of the components of the investigational product (including penicillin and streptomycin), or who can not receive treatment with antihistamines and/or corticosteroids.
4. Subjects with signs of active systemic infection at the time of inclusion in the study. In any case, according to the researcher's criteria, the patient can be reevaluated for inclusion in the study after improvement of the infectious pathology.
5. Subjects with a history or signs of malignancy, including cutaneous squamous cell carcinoma.
6. Subjects with circulating anti-C7 antibodies and anti-C7 antibodies deposited in the dermo-epidermal junction detected in skin biopsies by indirect immunofluorescence.
7. Pregnant women at the time of inclusion or women of childbearing age who do not practice abstinence or employ acceptable means of contraception, as determined by the investigator during the trial.
8. Biochemical abnormalities at the time of inclusion: albumin <2.5 g / dL, Hemoglobin <7.5 g / dL.
9. Subjects to whom other investigational drugs have been administered in the 90 days prior to the treatment phase.
10. Subjects who are unable to understand the information sheet and unable to sign the informed consent.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Incidence of Treatment-Emergent Adverse Events as assessed by protocol. | 1 year after infusion
  To evaluate the safety of haploidentical MSCs derived from bone marrow administered by intravenous injection with a dose of 2-3x106 cells / Kg in 3 infusions separated by 21 days each for the treatment of patients with RDEB: All adverse events will be registered for 1 year from first infusion of cells as assessed by grade: mild, moderate or severe (according to protocol)

SECONDARY OUTCOMES:
Cutaneous mechanical resistance | 2 year after infusion
  Cutaneous mechanical resistance measured using a negative pressure cutaneous suction device from Electronic Diversities (NP-2 model).
Skin surface affected | 2 year after infusion
  Percentage of skin surface affected in patients with RDEB
Number of blisters | 2 year after infusion
  Quantification of the number of blisters in patient with RDEB
Non-specific general markers of systemic inflammation: white blood cell count | 2 year after infusion
  Biomarkers evaluated are white blood cell count (109/L)
Non-specific general markers of systemic inflammation: Negative acute phase reactant (albumin) | 2 year after infusion
  Biomarkers evaluated are negative acute phase reactants: albumin (g/dl)
Non-specific general markers of systemic inflammation: Negative acute phase reactants (pre-albumin, transferrin and retinol-binding protein) | 2 year after infusion
  Biomarkers evaluated are negative acute phase reactants: pre-albumin, transferrin, and retinol-binding protein (mg/dl)
Non-specific general markers of systemic inflammation: Positive acute phase reactants (c-reactive protein and fibrinogen) | 2 year after infusion
  Biomarkers evaluated are positive acute phase reactants: C reactive protein and fibrinogen (mg/dl)
Non-specific general markers of systemic inflammation: Positive acute phase reactants (ferritin) | 2 year after infusion
  Biomarkers evaluated are positive acute phase reactants: ferritin (ng/ml)
Severity index according to "The Birmingham Epidermolysis Bullosa Severity Score" before and after treatment | 2 year after infusion
  The Birmingham Epidermolysis Bullosa Severity Score evaluated the severity of disease before and after treatment. Eleven items were scored: area of damaged skin, involvement of nails, mouth, eyes, larynx and oesophagus, scarring of hands, skin cancer, chronic wounds, alopecia and nutritional compromise (giving a maximum score of 100, where 0 = better outcome and 100 = worse outcome)
Severity index according to "The Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) before and after treatment | 2 year after infusion
  The Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) used to classify patients according to disease severity and clinical response in three types: mild, moderate and severe (obtained by the analysis of 12 skin sites in addition to the scalp, mucous membranes, nails and other epithelized surfaces - total activity (of 276) and damage (of 230) combine to give an overall score of 506; where 0 = better outcome and 506 = worse outcome).
Expression of Collagen VII (C7) in skin biopsy | 2 year after infusion
  Expression of Collagen VII (C7) in skin biopsy will be analyzed by immunofluorescence with antibodies specific for the NC1 domain of collagen VII.
Analysis of anchoring fibrils | 2 year after infusion
  Analysis of anchoring fibrils by electron microscopy in skin biopsy after treatment
Variation of pain respect to baseline status: Visual Analog Scale | 2 year after infusion
  Variation of pain with respect to baseline that will be assessed using the Visual Analogy Scale (VAS) in all visits after the first infusion, used different type of VAS scale depends on age of subject. Range was 1 to 10, where 10 are considered a worse outcome.
Modification in itching perceived | 2 year after infusion
  Assessment of the change in the itching perceived respect baseline status will be assessed by Leuven Itch Scale or Itch Man Scale, depends on the age of the subject. These scales are the instrument to evaluate itching perceived in patients with pruritus origin different. There subscale in 6 domains: frequency, duration, severity, distress, impact, and area: Itch frequency score: scale from 0 to 100. (Maximum score 100, itching all the time - is worse outcome) Itch severity score: scale from 0 to 100 (Maximum score 100, maximum severity =worse outcome) Itch distress score: scale from 0 to 100 (Maximum score 100, maximum distress = worse outcome) Itch consequences score: scale from 0 to 100 (Maximum score 100, maximum consequences = worse outcome) Itch Surface area score: Scale from 0 to 100 (Maximum score is 100, the entire body = worse outcome).
Change in quality of life of patient: European Quality of Life-5 Dimensions-5 level (EUROQL-5D) | 2 year after infusion
  Assessment of the change in quality of life: survey of specific assessment of the quality of life (European Quality of Life-5 Dimensions-5 level; EUROQL-5D). The descriptive system comprises five dimensions: mobility, self-care, habitual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of gravity, where a value of 1 is better outcome and 3 is worse outcome. Also, there are a 2nd part included a VAS scale, where 0 = worse outcome and 100 =better outcome.
Evaluation of circulating anti-C7 antibodies | 2 year after infusion
  Analysis of circulating anti-C7 antibodies determined by ELISA before and after treatment.
Change in general condition of the patient | 2 year after infusion
  Evaluation of the changes produced in the patient before and after the study treatment, assessing according to the set of tests performed on the patient during the same; indicating it through a Likert scale, from 1-4, where 4 is the most serious evaluation and 1 is the slightest.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain